CLINICAL TRIAL: NCT01603901
Title: Regulated Negative Pressure-Assisted Wound Therapy Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYMC-2012-31
Record Dates: First submitted 2012-05-20; First posted 2012-05-23 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Investigated Wounds (Experimental)
  Interventions: Device: Regulated Negative Pressure-Assisted Wound Therapy Device

INTERVENTIONS:
Device: Regulated Negative Pressure-Assisted Wound Therapy Device — Negative pressure will be applied in the usual way that is normally applied in our Medical Center

SUMMARY:
Regulated negative pressure-assisted wound therapy (RNPT) is regarded as a gold standard technology for treatment of various chronic and acute wounds. The investigators plan to evaluate the efficacy and ease of use of this device.

ELIGIBILITY:
Inclusion Criteria:

* Chronic or acute wounds

Exclusion Criteria:

* Uncontrolled bleeding
* Neoplasms in wound
* Exposed blood vessels
* Exposed internal organs

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-06; Primary Completion 2012-08 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy | Ten days
  Measurement of change in wound size

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel